CLINICAL TRIAL: NCT06865287
Title: Effects of a Tactical Critical Thinking Program on Tactical Efficiency in Elite Underwater Rugby Male Players
Acronym: TPCTUWR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Vicosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UWR Bioethical USB
Record Dates: First submitted 2025-02-21; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2023-09

CONDITIONS: Tactical Index; Critical Thinking Index
Keywords: Tactical Performance Index; Critical Thinking Index; Underwater Rugby; Socio-constructivist Approach

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization was performed using block random number generation [16], with block sizes of 4-6 and stratification based on experience (low: <2 years, medium: 2-4 years, high: >4 years). An external individual, independent of the research team, carried out the allocation to ensure unbiased group assignments. To minimize bias, participants were unaware of the study objectives or their group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard training routine (STR) group (Active Comparator): Both TPCT and STR groups will follow identical underwater rugby training sessions. Structure: Warm-up (15%): Land-based mobility (5 min) + in-water rondos (10 min). Small-Sided Games (30%): Tactical principles via modified scenarios. Full-Team Games (45%): 6v6, 5-min games with 3-min recovery. Cool-down (10%).
  Training includes 20 sessions: 8 defensive (Containment, Recovery) and 12 offensive (Penetration, Offensive Coverage, Space).
  SSGs focus on tactical principles:
  Containment (4v4, restricted defensive movement) → Defensive positioning, communication.
  Recovery (5v6, interception-based) → Quick transitions, passing accuracy. Penetration (4v2, lane-based) → Offensive coordination, defensive pressure. Offensive Coverage (6v6, restricted movement) → Off-the-ball play, passing options.
  Space (3v4, defenders in pairs) → Forward movement, spatial awareness.
  Interventions: Other: STR Group
- TPCT Group (Experimental): Both TPCT and STR groups followed identical underwater rugby training: Warm-up (15%), SSGs (30%), Full-Team Games (45%), Cool-down (10%). Training included 20 sessions: 8 defensive (Containment, Recovery) and 12 offensive (Penetration, Offensive Coverage, Space).
  SSGs focused on tactical principles:
  Containment (4v4) → Defensive positioning, communication. Recovery (5v6) → Quick transitions, passing accuracy. Penetration (4v2) → Offensive coordination, defensive pressure. Offensive Coverage (6v6) → Off-the-ball play, passing options. Space (3v4) → Forward movement, spatial awareness. The TPCT group engaged in 10-min reflective discussions post-warm-up, SSGs, and games. Prompts included: "What key moments defined the activity?" "How effective were our decisions?" "How well did we contain attackers?" "What hindered or helped recovery?" "How could we improve movement and space usage?" Players progressively led discussions, enhancing tactical awareness.
  Interventions: Other: TPCT Group

INTERVENTIONS:
Other: STR Group — Both TPCT and STR groups will follow identical underwater rugby training sessions. Structure: Warm-up (15%): Land-based mobility (5 min) + in-water rondos (10 min). Small-Sided Games (30%): Tactical principles via modified scenarios. Full-Team Games (45%): 6v6, 5-min games with 3-min recovery. Cool-down (10%).
  Training includes 20 sessions: 8 defensive (Containment, Recovery) and 12 offensive (Penetration, Offensive Coverage, Space).
  SSGs focus on tactical principles:
  Containment (4v4, restricted defensive movement) → Defensive positioning, communication.
  Recovery (5v6, interception-based) → Quick transitions, passing accuracy. Penetration (4v2, lane-based) → Offensive coordination, defensive pressure. Offensive Coverage (6v6, restricted movement) → Off-the-ball play, passing options.
  Space (3v4, defenders in pairs) → Forward movement, spatial awareness.
  Arms: Standard training routine (STR) group
Other: TPCT Group — Both TPCT and STR groups followed identical underwater rugby training: Warm-up (15%), SSGs (30%), Full-Team Games (45%), Cool-down (10%). Training included 20 sessions: 8 defensive (Containment, Recovery) and 12 offensive (Penetration, Offensive Coverage, Space).
  SSGs focused on tactical principles:
  Containment (4v4) → Defensive positioning, communication. Recovery (5v6) → Quick transitions, passing accuracy. Penetration (4v2) → Offensive coordination, defensive pressure. Offensive Coverage (6v6) → Off-the-ball play, passing options. Space (3v4) → Forward movement, spatial awareness. The TPCT group engaged in 10-min reflective discussions post-warm-up, SSGs, and games. Prompts included: "What key moments defined the activity?" "How effective were our decisions?" "How well did we contain attackers?" "What hindered or helped recovery?" "How could we improve movement and space usage?" Players progressively led discussions, enhancing tactical awareness.
  Arms: TPCT Group

SUMMARY:
The aim of this study was to examine the effects of the Tactical Programme for Critical Thinking (TPCT) on tactical performance and critical thinking (CT) skills in elite male underwater rugby (UWR) players. Twenty-four players (age: 29.38 ± 7.11 years; experience: 10.86 ± 4.82 years) were divided into two groups: one following a structured TPCT intervention and another maintaining their standard training routine (STR). The intervention consisted of 20 sessions (two per week) focused on tactical principles in UWR. Tactical performance was assessed using the RUSTAC test, while critical thinking skills were evaluated with the Critical Thinking Measurement Index.

DETAILED DESCRIPTION:
1. Introduction Performance in team sports relies heavily on effective decision-making in dynamic environments. The complexity of these settings, with constantly shifting variables, demands cognitive adaptability and problem-solving skills, moving beyond pre-set responses. Traditional coaching methods, often focusing on technique, can fall short in preparing athletes for the unpredictability of competition, hindering the development of problem-solving and adaptive decision-making. This is particularly true in sports like underwater rugby (UWR), where speed, precision, and creative thinking are essential.

   Tactical learning, integrating decision-making, problem-solving, and execution, offers a more holistic training approach. However, its effectiveness, especially for elite athletes, is debated, particularly regarding implicit vs. explicit learning. While implicit learning fosters adaptability, explicit methods provide structured guidance for mastering complex tactical behaviours. Research suggests elite athletes may benefit more from explicit, sport-specific training.

   The Tactical Programme for Critical Thinking (TPCT) offers a new approach to developing critical thinking and decision-making. Based on socio-constructivist theory, it emphasises active learning, reflection, and collaboration. Although initial TPCT applications in U-14 football have shown promise, its impact on elite athletes is less understood. Elite athletes may exhibit reduced sensitivity to training adaptations, but the TPCT's structured, explicit nature may be beneficial, particularly in complex sports like UWR, where tactical awareness is vital.

   This study evaluated the TPCT's effect on the Tactical Performance Index (TPI) and critical thinking (CT) in elite UWR players. By examining its impact in a high-performance setting, this research aimed to contribute to the understanding of explicit training methods and inform sports science and elite coaching practice.
2. Methods 2.1 Participants This study involved 27 elite male underwater rugby (UWR) players, all members of the reigning world club champions (August-October 2023). Participants were selected through a non-probabilistic method based on convenience and feasibility, ensuring the inclusion of world-class players.

   Players were classified as Tier 5 athletes, denoting world-class performance levels according to the Participant Classification Framework. This classification includes players ranked among the top 3-20 globally, finalists in World Championships, or those competing at the highest levels internationally. Notably, 14 of the 27 players were three-time world champions, underscoring the exceptional calibre of this cohort. The remaining players were multiple-time national champions with extensive elite-level experience, reinforcing the high expertise within the group.

   This study involved 24 elite male UWR players, divided into two groups: one following a structured Tactical Programme for Critical Thinking (TPCT) intervention and the other maintaining their standard training routine (STR). The TPCT group consisted of 11 players (M±SD: age = 30.84±7.20 years, experience = 10.50±6.41 years, height = 179.00±8.19 cm, mass = 87.83±11.90 kg), while the STR group included 13 players (M±SD: age = 28.28±7.88 years, experience = 11.12±3.28 years, height = 174.14±8.09 cm, mass = 85.94±12.80 kg). The intervention spanned 10 weeks, consisting of two training sessions per week, for a total of 20 sessions.

   The inclusion and exclusion criteria were carefully defined to ensure a reliable and homogeneous group of participants. Players had to meet the inclusion criteria both before and throughout the intervention. Specifically, they were required to maintain a minimum attendance rate of 80% during pre-intervention training sessions and demonstrate consistent commitment throughout the study. To enhance internal validity and minimise potential confounding variables, exclusion criteria were established. Players were excluded if they had musculoskeletal injuries or conditions that could impair their performance during the intervention. Additionally, those without medical clearance to participate in high-intensity underwater rugby sessions were not included. Engagement in other competitive team sports during the intervention period was also an exclusion factor, as it could introduce variability in physical and tactical adaptations. Furthermore, players with uncontrolled learning disorders or cognitive impairments that might interfere with their ability to understand and execute the intervention tasks effectively were excluded. These criteria were designed to ensure a sample of elite players who could fully adhere to the intervention protocol, reducing external influences that might confound the results. By addressing these potential confounders, the study aimed to provide a more accurate assessment of the intervention's effects on performance outcomes.

   Randomisation was performed using block random number generation, with block sizes of 4-6 and stratification based on experience (low: <2 years, medium: 2-4 years, high: >4 years). An external individual, independent of the research team, carried out the allocation to ensure unbiased group assignments. To minimise bias, participants were unaware of the study objectives or their group assignments.

   The intervention protocol was evaluated and approved by the bioethics committee of the local university on June 5, 2023. This study adhered to the principles outlined in the Declaration of Helsinki, ensuring the protection of participants' rights, dignity, and confidentiality throughout the research process. Informed consent was obtained from all participants, and they were fully briefed on the nature of the study, the voluntary nature of their involvement, and their right to withdraw at any time without penalty. All data collected were handled in accordance with ethical guidelines to ensure the participants' privacy and well-being. The study also complied with relevant national and international human rights regulations to ensure that the research was conducted in an ethical and responsible manner.

   2.2 Procedures This study was conducted at the Complejo Acuático de Medellín, Colombia, home of the Orcas Underwater Rugby Club.

   Timeline:

   Pre-testing: 7th - 11th August 2023 (Allow sufficient time for all assessments) Intervention: 14th August - 26th October 2023 (10 weeks, two sessions per week - Tuesdays and Thursdays) Post-testing: 29th October - 2nd November 2023 (Immediately following the intervention) Location:

   All training sessions and testing took place at the Complejo Acuático de Medellín, located at Medellín, Colombia. The pool dimensions are 12x18x5m and the water temperature is typically 28 degrees.

   Training Content:

   Both the TPCT and the standard training routine (STR) groups participated in identical underwater rugby training sessions, focusing on developing key tactical principles. The training sessions followed this structure:

   Warm-up (15%): Included land-based joint mobility exercises (5 minutes) followed by in-water rondos (10 minutes). Small-Sided Games (SSGs) with Tactical Manipulations (30%): Focused on specific tactical principles using modified game scenarios. Details of SSGs are provided below. Full-Team Games (6v6) (45%): 5-minute games with 3-minute recovery periods, allowing players to apply learned principles in a game context. Cool-down (10%): Light swimming and stretching. The 20 training sessions covered the following tactical principles with 8 sessions (40%) dedicated to defensive principles and 12 sessions (60%) focused on offensive principles:

   Session Range Tactical Principle Description Focus 1-4 Containment (Defensive) Stop or delay the opponent's attack. Positioning, communication, pressure. 5-8 Recovery (Defensive) Regain possession after losing the ball. Transition speed, counter-attacking. 9-12 Penetration (Offensive) Attack directly towards the opponent's goal. Speed, passing accuracy, support play. 13-16 Offensive Coverage (Offensive) Provide support to the ball carrier. Passing options, movement off the ball. 17-20 Space (Offensive) Use and expand the playing area. Width, depth, passing lanes.

   Detailed Small-Sided Game (SSG):

   Containment SSG (Sessions 1-4): Setup: Half-field (4m x 8m). 6v6 (3 attackers vs. 3 defenders per team). Rules: The attacking team (Team A) attempted to score by advancing the ball into the defensive zone. The defending team (Team B) contained the attack, with only two defenders allowed in their defensive half. Once Team A entered Team B's half, only two players from Team B actively defended; the remaining defenders stayed on the surface. If Team B recovered possession, all players from Team B joined the attack. If a goal was scored, the game restarted with all players. Players rotated between attacking and defending roles. Objectives: To develop defensive positioning, communication, and pressure to contain the attack and prevent scoring opportunities. To improve the ability of the surface players to quickly join the play when possession was regained. Focus: Defensive organisation, communication, quick transitions. Recovery SSG (Sessions 5-8): Setup: 3m x 8m playing area. 5v6 (5 attackers vs. 6 defenders). Rules: The attacking team (Team A) attempted to score. The defending team (Team B) could only intercept or block passes; they could not move with the ball. Team A players could not move with the ball; they passed to advance. If a goal was scored, the game restarted. Players rotated between attacking and defending roles.

   Objectives: To improve the defending team's ability to intercept passes and regain possession. To develop the attacking team's passing accuracy and ability to create scoring opportunities without moving with the ball. Focus: Interceptions, passing accuracy, quick reactions. Penetration SSG (Sessions 9-12): Setup: Half-field (4m x 8m) divided into two equal lanes (left and right). 4v2 (4 attackers vs. 2 defenders). Rules: The attacking team (Team A) started with the ball and attacked within their designated lane. Only two players from Team A were allowed in each lane. Defenders (Team B) moved freely. If Team A lost possession, two players from Team B entered the field, two players from Team A left, and the roles reversed. Objectives: To develop attacking players' ability to penetrate the defence using lane discipline and coordinated movements. To improve defenders' ability to defend against attacks in confined spaces. Focus: Attacking in lanes, defensive pressure. Offensive Coverage SSG (Sessions 13-16): Setup: Half-field (4m x 8m). 6v6 (attackers vs. defenders). Rules: The attacking team (Team A) started with the ball. Attacking players moved without the ball. Defending players (Team B) were positioned strategically in their defensive zone and did not move; they intercepted the ball from their position. If Team A lost possession, they regained it and continued the attack. Objectives: To develop attacking players' off-the-ball movement and ability to create passing options. To improve defenders' ability to read the attack and intercept passes from static positions. Focus: Movement off the ball, passing options, defensive positioning. Space SSG (Sessions 17-20): Setup: Half-field (4m x 8m). 3v4 (3 attackers vs. 4 defenders). Rules: The attacking team (Team A) started with the ball and moved forwards. The defending team (Team B) worked in two pairs; each pair held hands and moved as a unit. Defenders intercepted from their combined position. If Team A lost possession, roles reversed. Objectives: To develop attacking players' ability to create and utilise space through forward movement. To improve defenders' ability to defend as a unit and intercept passes. Focus: Forward movement, creating space, coordinated defence. TPCT Specifics (TPCT Group): The TPCT group engaged in structured reflective discussions after the warm-up, after the SSGs, and after the full-team games. These discussions were facilitated by the coach and lasted approximately 10 minutes each. The coach guided the discussions using open-ended questions and prompts designed to encourage critical thinking and reflection on tactical decision-making. Prompts: General: "What were the key moments in that activity?" "How effective were tactical decisions?" "What could have been done differently?" Containment: "How well were the attackers contained?" "What communication strategies were most effective?" Recovery: "How quickly was the transition from defence to attack?" "What factors hindered or helped recovery efforts?" Penetration: "How successful were penetration attempts?" "What passing strategies created the best scoring opportunities?" Offensive Coverage: "Was adequate support provided to the ball carrier?" "How could movement off the ball be improved?" Space: "Was the available space effectively utilised?" "How can more passing lanes be created?" The coach encouraged players to analyse their performance, identify areas for improvement, and develop strategies for future actions. The reflection process evolved over the 10 weeks, with players gradually taking more ownership of the discussions. STR Group Activities: The STR group followed the same training content as the TPCT group, but did not participate in structured reflective discussions. During the periods when the TPCT group was reflecting, the STR group rested, hydrated, and received general feedback from the coaching staff. Free Play: In addition to the structured training sessions, both groups participated in free play scrimmages 2 times per week, for a duration of 40 minutes each time. These scrimmages simulated real-game conditions, allowing players to apply learned tactical principles in a dynamic and unpredictable environment. No formal reflection took place during or after free play. Standardisation of Pre- and Post-Test Conditions: To ensure the reliability of pre- and post-test assessments, the following measures were implemented: Participants refrained from high-intensity training, caffeine intake, and cognitively demanding activities for 48 hours prior to testing to minimise fatigue-related confounding factors. Pilot testing was conducted to optimise camera placement, action counting, and data processing protocols, ensuring methodological rigor. Video analysts received detailed training in data analysis, following specific guidelines for the test methodology. Strict adherence to player selection criteria was maintained, with thorough verification to ensure data integrity. Pilot tests focused on refining camera placement, action counting, and data coding, addressing any issues before full-scale implementation. Data Collection Procedures: Data was collected using waterproof digital cameras (GoPro Hero 5) with a resolution of 1080p and a frame rate of 120 FPS. This setup captured high-quality footage of training sessions and scrimmages. The camera operator performed panning movements to actively track the ball and key player movements, providing continuous coverage of the game for RUSTAC coding. Prior to the study, all equipment was calibrated and tested. Evaluators underwent a two-stage training protocol: Theoretical Training: Evaluators were trained on the use of the RUSTAC tool, including a written assessment to confirm understanding. Practical Training: Evaluators analysed game sequences from pilot test footage, with feedback sessions to refine accuracy and consistency. Inter-rater reliability (Cohen's Kappa) and intra-observer reliability (Cohen's Kappa) were assessed to ensure the reliability of the evaluation process. 2.6 Instruments Tactical Performance Assessment: Tactical performance was assessed using the validated RUSTAC instrument (Content Validity Coefficient: 0.92). RUSTAC provides a comprehensive framework for evaluating tactical actions in underwater rugby, focusing on offensive and defensive principles. Five key variables were assessed: penetration, offensive coverage, space, defensive coverage, and recovery. Tactical Performance Indices (TPI) were calculated for offensive and defensive zones, along with a general gameplay efficiency index. Field Test Setup: 3v3 scrimmages were conducted on an 8m x 6m field, adhering to RUSTAC methodology. Each scrimmage consisted of two 90-second periods separated by a 60-second recovery interval. Players from the TPCT and STR groups were mixed and assigned to alternating teams (blue and white gear) to ensure balanced skill levels. A standardised warm-up, consisting of 100m swimming without fins and 200m with fins at low intensity, was performed before each test. The playing field was divided into offensive and defensive zones to facilitate observation of transitions. An offensive sequence was defined as beginning with ball possession and the team actively attempting to advance towards the opponent's goal/basket, concluding when possession was lost or a goal was scored. Tactical Performance Calculation: All actions were coded according to the RUSTAC categories (Table 1). Effectiveness was evaluated, and TPIs were calculated as the ratio of successful actions to total actions, expressed per 100 actions. Full details of the RUSTAC coding system, area dimensions, scrimmage durations, and TPI calculation methodology are available in the original publication. Table 1 (below) provides a summary of the tactical principles assessed. Table 1. Tactical principles in underwater rugby Offensive Phase with Ball Possession Defensive Phase without Ball Possession Penetration Containment and Concentration Attack (with ball possession) directly to the end line or the basket. Stop or delay the opponent's attack or counterattack. Offensive Coverage Defensive Coverage Provide support to the ball carrier by offering passing options for the continuation of the play. Serve as an additional obstacle to the ball carrier if they pass the ball. Space Recovery Use and expand the effective playing space of the team by ensuring passing lines. Allow the team to recover the ball in any play area. Mobility and Offensive Unity Create passing lines in depth during defence-to-offense transitions.

   Critical Thinking Assessment:

   Critical thinking (CT) was assessed using the IMPC OSBA VS2 (Critical Thinking Measurement Index VS2), developed in Medellín, Colombia. This instrument evaluates CT based on competencies including evaluation, argumentation, analysis, inference, and interpretation. Although designed for higher education students, the instrument was adapted for this study's participants (also from Medellín) to ensure cultural relevance and compatibility. The instrument's reliability was established with a Cronbach's alpha of 0.659, demonstrating acceptable internal consistency. Validity was confirmed via the Kaiser-Meyer-Olkin (KMO) test (0.52) and Bartlett's test (p < 0.001). The instrument explains 69.48% of the variance, indicating its capacity to effectively assess key CT dimensions.

   Participant responses were scored following the original authors' methodology. Raw scores derived from participant answers were used to calculate final CT scores. As access to the original developers' data is unavailable, the scoring methodology outlined in the original validation work was strictly adhered to in this study.

   2.7 Data Collection Data was collected using waterproof digital cameras (GoPro Hero 5) with a resolution of 1080p and a frame rate of 120 FPS. Video recordings were made of all training sessions, including warm-ups, small-sided games, full-team games, and free play scrimmages. Cameras were positioned to provide a comprehensive view of the playing field, with panning to follow the flow of play and capture all relevant tactical actions. Specific camera placements included overhead view and sideline view. Recording protocols ensured consistent lighting.

   2.8 Data Analysis Data analysis was performed using SPSS software (Version 25; IBM Corp, Armonk, NY, USA) and GraphPad Prism (Version 5; GraphPad Software, San Diego, CA, USA) for data visualisation.

   Prior to analysis, data normality was assessed using the Shapiro-Wilk test for datasets with fewer than 50 data points. Levene's test was used to assess the homogeneity of variances. Descriptive statistics were presented as means and standard deviations for normally distributed variables, and as medians and interquartile ranges for non-normally distributed variables.

   To compare pre- and post-intervention data between the TPCT and STR groups, independent samples t-tests were used for normally distributed variables, and Mann-Whitney U tests were used for non-normally distributed variables. Intragroup differences were also assessed, and percentage changes were calculated as: ((post-intervention value - pre-intervention value) / pre-intervention value) * 100.

   Effect sizes were calculated to determine the magnitude of observed differences. Cohen's d was used for parametric data, and the rank-biserial correlation coefficient was used for non-parametric data. Cohen's d effect sizes were interpreted as small (0.2), medium (0.5), and large (0.8). Rank-biserial correlation effect sizes were interpreted as small (0.1), medium (0.3), and large (0.5). The alpha level for statistical significance was set at (Specify alpha level, usually 0.05).
3. Ethical Considerations Ethical approval was obtained from the Ethics Committee at Universidad San Buenaventura, Medellín Colombia before the study commenced. The study adhered to the Declaration of Helsinki. All participants provided written informed consent after receiving a full explanation of the study's purpose, procedures, risks, and benefits. Participants were free to withdraw from the study at any time without penalty.

ELIGIBILITY:
Inclusion Criteria:

* 24 elite male underwater rugby (UWR) players.
* Members of the reigning world club champions (August-October 2023).
* Selected via a non-probabilistic method based on convenience and feasibility.
* Required to have no musculoskeletal injuries at the start of the study.
* Maintained a minimum attendance rate of 80% during pre-intervention training sessions.
* Demonstrated consistent commitment throughout the study.

Exclusion Criteria:

* Active musculoskeletal injuries at the start of the study that could affect performance.
* Recent history of surgery or severe injuries within the past six months.
* Attendance below 80% in pre-intervention training sessions.
* Lack of commitment to the study, demonstrated by low engagement or inconsistent participation in training.
* Pre-existing medical conditions that could limit participation in high-intensity activities.
* Insufficient competitive experience, meaning players without prior participation in high-level tournaments.
* Use of prohibited substances or doping methods as per current sports regulations.
* Simultaneous participation in another training programme, which could interfere with the study's intervention.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Tactical Efficiency Index | Week one and Ten
  Description: Data analysis in this study utilised the Tactical Underwater Rugby Test (RUSTAC) instrument, which has been validated for use in underwater rugby (Content Validity Coefficient: 0.92). RUSTAC provides a comprehensive evaluation of tactical actions in gameplay, focusing on key principles of offensive and defensive phases. The instrument was used to assess five key variables during gameplay: penetration, offensive coverage, space, defensive coverage, and recovery. Additionally, Tactical Performance Indices (TPI) were calculated for both offensive and defensive zones, and general gameplay efficiency. The Tactical Performance Indices are scored on a scale from 0 to 1, where 1 indicates the highest efficiency and 0 the lowest efficiency. Therefore, higher scores represent better tactical performance.
Critical Thinking | Week one and Ten
  Critical thinking was assessed using the IMPC OSBA VS2 (Critical Thinking Measurement Index VS2), developed in Medellín, Colombia. This instrument evaluates critical thinking via evaluation, argumentation, analysis, inference, and interpretation. Adapted for participants from Medellín, it ensures cultural relevance. Reliability (Cronbach's alpha 0.659) and validity (KMO 0.52, Bartlett's p<0.001) were confirmed. It explains 69.48% of variance. Scored 0-100, 100 is highest critical thinking; higher scores indicate better skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Antioquia Institute of Technology, Medellín, Colombia

IPD SHARING:
Plan to Share IPD: No